CLINICAL TRIAL: NCT02954393
Title: Influence of Moment of Systemic Metronidazole and Amoxicillin Administration in the Treatment of Chronic Periodontitis: a Randomized Clinical Trial.
Brief Title: Amoxicillin and Metronidazole During Periodontal Treatment
Acronym: MOMENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Belén Retamal-Valdes (Other)
Responsible Party: Sponsor-Investigator, Belén Retamal-Valdes, DDS, MSc, PhD Student, University of Guarulhos
Organization: University of Guarulhos (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE: 32465714.4.1001.5506
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Chronic Periodontitis
Keywords: Periodontal disease; Metronidazole; Amoxicillin; Scaling and root planing; Healing phase
MeSH Terms: conditions — Chronic Periodontitis; Periodontal Diseases | interventions — Tooth Exfoliation; Root Planing; P-2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Scaling and root planing + Placebos active phase thrice a day (TID) for 14 days and Placebos healing phase TID for 14 days.
  Interventions: Procedure: Scaling and root planing; Drug: Placebos active phase; Drug: Placebos healing phase
- Active phase (Active Comparator): Scaling and root planing + Metronidazole active phase (400 mg/thrice a day,TID) + Amoxicillin active phase (500 mg/ TID) for 14 days and Placebos healing phase TID for 14 days.
  Interventions: Procedure: Scaling and root planing; Drug: Metronidazole active phase; Drug: Amoxicillin active phase; Drug: Placebos healing phase
- Healing phase (Active Comparator): Scaling and root planing + Placebos active phase thrice a day (TID) for 14 days and Metronidazole healing phase (400 mg/TID) + Amoxicillin healing phase (500 mg/TID) for 14 days.
  Interventions: Procedure: Scaling and root planing; Drug: Metronidazole healing phase; Drug: Amoxicillin healing phase; Drug: Placebos active phase

INTERVENTIONS:
Procedure: Scaling and root planing — SRP will be performed in four to six appointments lasting approximately 1 h each, using manual curettes (Hu-Friedy, Chicago, IL, USA) and ultrasonic device (Cavitron Select SPC, Dentsply professional, York, PA, USA) under local anesthesia. The deep sites will be scaled throughout the first week and treatment of the entire oral cavity will be completed in 14 days.
  Other Names: SRP
Drug: Metronidazole active phase — Metronidazole 400 mg thrice a day for 14 days in the active phase of the periodontal treatment (beginning with the first SRP session).
  Other Names: MTZ 1
  Arms: Active phase
Drug: Metronidazole healing phase — Metronidazole 400 mg thrice a day for 14 days in the healing phase of the periodontal treatment (3 months after active phase).
  Other Names: MTZ 2
  Arms: Healing phase
Drug: Amoxicillin active phase — Amoxicillin 500 mg thrice a day for 14 days in the active phase of the periodontal treatment (beginning with the first SRP session).
  Other Names: AMX 1
  Arms: Active phase
Drug: Amoxicillin healing phase — Amoxicillin 500 mg thrice a day for 14 days in the healing phase of the periodontal treatment (3 months after active phase).
  Other Names: AMX 2
  Arms: Healing phase
Drug: Placebos active phase — Amoxicillin and metronidazole placebos thrice a day for 14 days in the active phase (beginning with the first SRP session).
  Other Names: P 1
  Arms: Control; Healing phase
Drug: Placebos healing phase — Amoxicillin and metronidazole placebos thrice a day for 14 days in the healing phase (3 months after active phase).
  Other Names: P 2
  Arms: Active phase; Control

SUMMARY:
The aim of this multicenter randomized clinical trial is to compare the clinical, microbiological and immunological effects of the adjunctive use of systemic metronidazole plus amoxicillin administered in different phases of the treatment of generalized chronic periodontitis.

DETAILED DESCRIPTION:
The combination of systemic metronidazole (MTZ) and amoxicillin (AMX) to scaling and root planing (SRP) has shown to be a promising periodontal treatment. However, some essential issues associated with the use of these antibiotics remain to be established. Although these agents are often prescribed after the healing phase of the SRP procedure, there is biological plausibility to support its use in conjunction with the mechanical treatment. However, to date, no placebo controlled randomized clinical trial (RCT) has directly compared these two protocols. Therefore, the aim of this multicentric RCT is to compare the clinical, microbiological and immunological effects of adjunctive systemic MTZ+AMX administered in different phases of the treatment of generalized chronic periodontitis (GChP). 180 subjects with GChP will be randomly assigned into three groups (n=60/group) that will receive SRP-only (control group) or in combination with 400 mg MTZ+500 mg AMX beginning at the first SRP session (group test 1) or after 3 months of its completion (group test 2). All volunteers will receive clinical and microbiological evaluation at baseline, 3, 6 and 12 months, and immunological assessment (levels of 20 chemokines) at baseline and 12 months post-therapy. Nine subgingival biofilm samples will be collected by subject and analyzed for counts and proportions of 40 bacterial species by checkerboard DNA-DNA hybridization. Differences in clinical, microbiological and immunological parameters among groups and over time will be evaluated using the ANOVA, ANCOVA, Chi-square and Tukey tests. Microbiological analyzes will be performed using adjustments for multiple comparisons. Statistical significance will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* ≥35 years of age;
* at least 15 teeth (excluding third molars and teeth with advanced decay indicated for extraction);
* a minimum of 6 teeth with at least one site each with probing depth (PD) and clinical attachment level (CAL) ≥5 mm;
* at least 30% of the sites with PD and CAL ≥4 mm and bleeding on probing (BOP).

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* current smoking and former smoking within the past 5 years;
* systemic diseases that could affect the progression of periodontitis (e.g. diabetes, immunological disorders, osteoporosis);
* scaling and root planing an in the previous 6 months;
* antibiotic therapy in the previous 6 months;
* long-term intake of anti-inflammatory medications;
* need for antibiotic pre-medication for routine dental therapy;
* use of orthodontic appliances;
* extensive dental prosthetic rehabilitation;
* allergy to metronidazole and/or amoxicillin.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-05; Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects reaching ≤ 4 periodontal sites with probing depth (PD) ≥ 5 mm at 12 months | 12 months

SECONDARY OUTCOMES:
Number of sites with PD ≥ 5 mm. | Baseline, 3, 6 and 12 months.
Number of sites with PD ≥ 6 mm. | Baseline, 3, 6 and 12 months.
Number of sites with PD ≥ 7 mm. | Baseline, 3, 6 and 12 months.
Reduction in the number of sites with PD ≥ 5 mm. | Baseline, 3, 6 and 12 months.
Reduction in the number of sites with PD ≥ 6 mm. | Baseline, 3, 6 and 12 months.
Reduction in the number of sites with PD ≥ 7 mm. | Baseline, 3, 6 and 12 months.
Mean PD changes in sites with initial PD between 4-6 mm | Baseline - 12 months.
Mean PD changes in sites with initial PD ≥ 7 mm. | Baseline - 12 months.
Mean CAL changes in sites with initial CAL between 4-6 mm | Baseline - 12 months.
Mean CAL changes in sites with initial CAL ≥ 7 mm. | Baseline - 12 months.
Full-mouth PD. | Baseline, 3, 6 and 12 months.
Full-mouth clinical attachment level. | Baseline, 3, 6 and 12 months.
Percentage of sites with bleeding on probing. | Baseline, 3, 6 and 12 months.
Percentage of sites with plaque accumulation | Baseline, 3, 6 and 12 months.
Percentage of sites with marginal bleeding. | Baseline, 3, 6 and 12 months.
Occurrence of headache obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of vomiting obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of diarrhea obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of metallic taste obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of nausea obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of irritability obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Proportions of periodontal pathogenic bacterial species. | Baseline, 3, 6 and 12 months.
Counts of periodontal pathogenic bacterial species. | Baseline, 3, 6 and 12 months.
Counts of chemokines in the crevicular gingival fluid. | Baseline and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Magda Feres, Professor, Study Chair — University of Guarulhos
Locations (2):
- Brazil (2):
  - University of Guarulhos, Guarulhos, São Paulo
  - University of São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] Feres M, Soares GM, Mendes JA, Silva MP, Faveri M, Teles R, Socransky SS, Figueiredo LC. Metronidazole alone or with amoxicillin as adjuncts to non-surgical treatment of chronic periodontitis: a 1-year double-blinded, placebo-controlled, randomized clinical trial. J Clin Periodontol. 2012 Dec;39(12):1149-58. doi: 10.1111/jcpe.12004. Epub 2012 Sep 27. PMID 23016867
- [Background] Feres M, Figueiredo LC, Soares GM, Faveri M. Systemic antibiotics in the treatment of periodontitis. Periodontol 2000. 2015 Feb;67(1):131-86. doi: 10.1111/prd.12075. PMID 25494600
- [Background] Haffajee AD, Patel M, Socransky SS. Microbiological changes associated with four different periodontal therapies for the treatment of chronic periodontitis. Oral Microbiol Immunol. 2008 Apr;23(2):148-57. doi: 10.1111/j.1399-302X.2007.00403.x. PMID 18279183
- [Background] Herrera D, Sanz M, Jepsen S, Needleman I, Roldan S. A systematic review on the effect of systemic antimicrobials as an adjunct to scaling and root planing in periodontitis patients. J Clin Periodontol. 2002;29 Suppl 3:136-59; discussion 160-2. doi: 10.1034/j.1600-051x.29.s3.8.x. PMID 12787214
- [Background] Keestra JA, Grosjean I, Coucke W, Quirynen M, Teughels W. Non-surgical periodontal therapy with systemic antibiotics in patients with untreated chronic periodontitis: a systematic review and meta-analysis. J Periodontal Res. 2015 Jun;50(3):294-314. doi: 10.1111/jre.12221. Epub 2014 Aug 21. PMID 25142259
- [Background] Lang NP, Tonetti MS. Periodontal risk assessment (PRA) for patients in supportive periodontal therapy (SPT). Oral Health Prev Dent. 2003;1(1):7-16. PMID 15643744
- [Background] Matuliene G, Pjetursson BE, Salvi GE, Schmidlin K, Bragger U, Zwahlen M, Lang NP. Influence of residual pockets on progression of periodontitis and tooth loss: results after 11 years of maintenance. J Clin Periodontol. 2008 Aug;35(8):685-95. doi: 10.1111/j.1600-051X.2008.01245.x. Epub 2008 Jul 23. PMID 18549447
- [Background] Matuliene G, Studer R, Lang NP, Schmidlin K, Pjetursson BE, Salvi GE, Bragger U, Zwahlen M. Significance of Periodontal Risk Assessment in the recurrence of periodontitis and tooth loss. J Clin Periodontol. 2010 Feb;37(2):191-9. doi: 10.1111/j.1600-051X.2009.01508.x. Epub 2009 Dec 21. PMID 20041980
- [Background] Mestnik MJ, Feres M, Figueiredo LC, Duarte PM, Lira EA, Faveri M. Short-term benefits of the adjunctive use of metronidazole plus amoxicillin in the microbial profile and in the clinical parameters of subjects with generalized aggressive periodontitis. J Clin Periodontol. 2010 Apr;37(4):353-65. doi: 10.1111/j.1600-051X.2010.01538.x. PMID 20447259
- [Background] Mestnik MJ, Feres M, Figueiredo LC, Soares G, Teles RP, Fermiano D, Duarte PM, Faveri M. The effects of adjunctive metronidazole plus amoxicillin in the treatment of generalized aggressive periodontitis: a 1-year double-blinded, placebo-controlled, randomized clinical trial. J Clin Periodontol. 2012 Oct;39(10):955-61. doi: 10.1111/j.1600-051X.2012.01932.x. Epub 2012 Aug 6. PMID 22882646
- [Background] Sgolastra F, Gatto R, Petrucci A, Monaco A. Effectiveness of systemic amoxicillin/metronidazole as adjunctive therapy to scaling and root planing in the treatment of chronic periodontitis: a systematic review and meta-analysis. J Periodontol. 2012 Oct;83(10):1257-69. doi: 10.1902/jop.2012.110625. Epub 2012 Feb 14. PMID 22220767
- [Background] Socransky SS, Haffajee AD. Dental biofilms: difficult therapeutic targets. Periodontol 2000. 2002;28:12-55. doi: 10.1034/j.1600-0757.2002.280102.x. No abstract available. PMID 12013340
- [Background] Socransky SS, Haffajee AD. Periodontal microbial ecology. Periodontol 2000. 2005;38:135-87. doi: 10.1111/j.1600-0757.2005.00107.x. No abstract available. PMID 15853940
- [Background] Socransky SS, Haffajee AD, Cugini MA, Smith C, Kent RL Jr. Microbial complexes in subgingival plaque. J Clin Periodontol. 1998 Feb;25(2):134-44. doi: 10.1111/j.1600-051x.1998.tb02419.x. PMID 9495612
- [Background] Socransky SS, Haffajee AD, Smith C, Dibart S. Relation of counts of microbial species to clinical status at the sampled site. J Clin Periodontol. 1991 Nov;18(10):766-75. doi: 10.1111/j.1600-051x.1991.tb00070.x. PMID 1661305
- [Background] Socransky SS, Smith C, Martin L, Paster BJ, Dewhirst FE, Levin AE. "Checkerboard" DNA-DNA hybridization. Biotechniques. 1994 Oct;17(4):788-92. PMID 7833043
- [Background] Teles RP, Haffajee AD, Socransky SS. Microbiological goals of periodontal therapy. Periodontol 2000. 2006;42:180-218. doi: 10.1111/j.1600-0757.2006.00192.x. No abstract available. PMID 16930311
- [Derived] Khattri S, Kumbargere Nagraj S, Arora A, Eachempati P, Kusum CK, Bhat KG, Johnson TM, Lodi G. Adjunctive systemic antimicrobials for the non-surgical treatment of periodontitis. Cochrane Database Syst Rev. 2020 Nov 16;11(11):CD012568. doi: 10.1002/14651858.CD012568.pub2. PMID 33197289
- [Derived] Feres M, Retamal-Valdes B, Mestnik MJ, de Figueiredo LC, Faveri M, Duarte PM, Fritoli A, Faustino E, Souto MLS, de Franco Rodrigues M, Giudicissi M, Nogueira BCL, Saraiva L, Romito GA, Pannuti CM. The ideal time of systemic metronidazole and amoxicillin administration in the treatment of severe periodontitis: study protocol for a randomized controlled trial. Trials. 2018 Mar 27;19(1):201. doi: 10.1186/s13063-018-2540-8. PMID 29587808